CLINICAL TRIAL: NCT04798391
Title: Effectiveness of Dexamethasone With Lignocaine for Alleviation of Tinnitus
Brief Title: Effectiveness of Intratympanic Dexamethasone With Ligmocaine for Alleviation of Tinnitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Combined Military Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, FARAH AFZAL, CLASSIFIED SPECIALIST, Combined Military Hospital, Pakistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMHQ
Record Dates: First submitted 2021-03-06; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Dexamethasone; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dexamethasone with lignocaine (Experimental)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Steroids and analgesics
  Other Names: Lignocaine

SUMMARY:
Objective: To determine the effectiveness of Intratympanic dexamethasone with lignocaine in control of idiopathic tinnitus.

Methodology: 264 consenting patients with idiopathic unilateral tinnitus presenting at ENT Department were assessed for tinnitus severity using Modified Tinnitus Handicap Inventory and the scores recorded and subsequently administered intratympanically 2.0 ml (milliliter's) of dexamethasone and lignocaine (1.5 ml dexamethasone + 0.5 ml 1% lignocaine). The dose was repeated twice at weekly intervals. All patients were re assessed on Modified Tinnitus Handicap Inventory two weeks after third Intratympanic administration.

ELIGIBILITY:
Inclusion Criteria:

* score 20 or above on modified tinnitus handicap inventory

Exclusion Criteria:

* head trauma, tympanic membrane perforation, depression, ear surgery

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Tinnitus relief | 2 weeks
  Tinnitus relief ascertained by Modified Tinnitus Handicap Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Combined Military Hospital, Quetta, Balochistan, Pakistan

IPD SHARING:
Plan to Share IPD: No